CLINICAL TRIAL: NCT07061249
Title: Effects of a 12-Week Waltz Dance Intervention on Cardiovascular Health in Women Aged 45-65 With Dyslipidemia: A Randomized Controlled Trial
Brief Title: Effects of a 12-Week Waltz Dance Intervention on Cardiovascular Health in Women Aged 45-65 With Dyslipidemia
Acronym: WD&CWD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gdansk University of Physical Education and Sport (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AWFiS/2025_5_JL
Record Dates: First submitted 2025-06-23; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Dyslipidemia; Cardiopulmonary Fitness
Keywords: Waltz Dance; Cardiopulmonary Fitness; Lipid Metabolism; Non-pharmacological Intervention; Aging
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Participants in this arm will receive a structured Waltz dance intervention as moderate-intensity aerobic exercise. The program consists of 3 supervised sessions per week for 12 weeks, each lasting 105 minutes. Each session includes a 5-minute warm-up, 50 minutes of solo and partner Waltz practice, a 5-minute rest, 40 minutes of choreographed combinations, and a 5-minute cool-down. The dance routines are progressive and designed to improve cardiovascular fitness, coordination, and balance. Exercise intensity is maintained at 50-70% of estimated maximum heart rate, with music tempo and movement complexity adjusted as needed. Physical activity is monitored using accelerometers to ensure target intensity is achieved.
  Interventions: Behavioral: Waltz Dance
- Control group (No Intervention): Only daily activities are included.

INTERVENTIONS:
Behavioral: Waltz Dance — Participants in this arm will receive a structured Waltz dance intervention as moderate-intensity aerobic exercise. The program consists of 3 supervised sessions per week for 12 weeks, each lasting 105 minutes. Each session includes a 5-minute warm-up, 50 minutes of solo and partner Waltz practice, a 5-minute rest, 40 minutes of choreographed combinations, and a 5-minute cool-down. The dance routines are progressive and designed to improve cardiovascular fitness, coordination, and balance. Exercise intensity is maintained at 50-70% of estimated maximum heart rate, with music tempo and movement complexity adjusted as needed. Physical activity is monitored using accelerometers to ensure target intensity is achieved.
  Arms: Exercise group

SUMMARY:
The goal of this clinical trial is to learn whether Waltz dance can improve cardiometabolic and bone health in sedentary women aged 45-65 with abnormal lipid levels. The main questions it aims to answer are:

Can Waltz dance improve blood lipid profiles, including total cholesterol, triglycerides, HDL-C, and LDL-C? Can it improve body composition, cardiorespiratory fitness, vascular function, and bone mineral density? Researchers will compare a Waltz dance group with a control group that maintains their usual lifestyle to see if the dance intervention leads to better health outcomes.

Participants will:

Attend supervised Waltz dance classes three times a week for 12 weeks, each session lasting 105 minutes.

Complete physical tests and blood draws before and after the program to measure changes in lipid levels, body composition, fitness, and bone density.

Wear an accelerometer to monitor energy expenditure and physical activity during the program.

ELIGIBILITY:
Inclusion Criteria:

1. Female participants aged between 45 and 65 years.
2. Diagnosed with dyslipidemia (based on clinical lipid profile: TC ≥ 6.2 mmol/L, TG ≥ 2.3 mmol/L, LDL-C ≥ 4.1 mmol/L, or HDL-C < 1.0 mmol/L).
3. Sedentary lifestyle (less than 60 minutes of structured physical activity per week in the last 6 months).
4. Able to participate safely in moderate-intensity exercise as confirmed by a medical evaluation.
5. Willing to participate in a 12-week supervised exercise program, 3 times per week.
6. Able to understand study procedures and provide written informed consent.

Exclusion Criteria:

1. Diagnosis of cardiovascular disease requiring medical supervision during exercise (e.g., unstable angina, recent myocardial infarction).
2. Severe musculoskeletal disorders (e.g., advanced osteoarthritis, recent fractures) limiting mobility or physical activity.
3. Neurological or cognitive disorders affecting motor function or communication.
4. Uncontrolled hypertension (SBP ≥ 160 mmHg or DBP ≥ 100 mmHg at rest).
5. Diagnosed osteoporosis with high fracture risk (T-score ≤ -2.5 and history of fragility fractures).
6. Any endocrine disorder that significantly affects lipid metabolism (e.g., uncontrolled thyroid disease, Cushing's syndrome).
7. Participation in structured exercise or dance programs within the past 12 months.
8. Current use of medications significantly affecting lipid levels (e.g., high-dose statins) unless dose has been stable for at least 3 months.
9. Any condition judged by the investigator to interfere with safe participation in the study.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-07-05 (Estimated); Primary Completion 2025-10-05 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Total Cholesterol (TC) Level | From enrollment to the end of treatment at 12 weeks
  Total cholesterol (TC) levels will be measured using fasting venous blood samples collected at baseline and after 12 weeks of intervention. Blood will be drawn in the morning after at least 8 hours of fasting. Serum will be analyzed in a certified laboratory using standard enzymatic colorimetric assays. TC is expressed in milligrams per deciliter (mg/dL). Elevated TC is a known risk factor for cardiovascular disease. Changes from baseline to post-intervention will be calculated.
Triglycerides (TG) Level | From enrollment to the end of treatment at 12 weeks
  Triglyceride (TG) levels will be assessed through fasting blood samples taken before and after the 12-week intervention. Samples will be processed using standardized laboratory techniques. TG is measured in mg/dL and high levels are associated with increased risk for metabolic and cardiovascular conditions. This outcome measures the change in TG levels between baseline and the end of the study.
High-Density Lipoprotein Cholesterol (HDL-C) Level | From enrollment to the end of treatment at 12 weeks
  HDL-C will be measured in serum obtained from fasting venous blood samples collected at baseline and 12 weeks. HDL-C is commonly known as "good" cholesterol due to its protective effect against cardiovascular disease. Standard enzymatic methods will be used for quantification. The change in HDL-C from baseline to post-intervention will be analyzed.
Low-Density Lipoprotein Cholesterol (LDL-C) Level | From enrollment to the end of treatment at 12 weeks
  LDL-C will be measured from fasting blood samples collected at the beginning and end of the 12-week intervention. LDL-C, often referred to as "bad" cholesterol, is a key risk factor for atherosclerosis and cardiovascular disease. The value will be determined using direct measurement or calculation by the Friedewald formula. Results will be reported in mg/dL, and changes from baseline to week 12 will be evaluated.

SECONDARY OUTCOMES:
Systolic and Diastolic Blood Pressure and Pulse Pressure (mmHg) | From enrollment to the end of treatment at 12 weeks
  Resting systolic blood pressure (SBP), diastolic blood pressure (DBP), and pulse pressure (PP = SBP - DBP) will be measured using an automated upper-arm blood pressure monitor (e.g., Omron HEM-7136). Participants will rest quietly in a seated position for at least 5 minutes before three measurements are taken on the right arm. The average of the three readings will be recorded.
Pulse Wave Velocity (m/s) | From enrollment to the end of treatment at 12 weeks
  Carotid-femoral pulse wave velocity (cfPWV), an indicator of arterial stiffness and vascular function, will be measured using a validated device (e.g., Complior Analyse). Measurements will be taken while participants are in the supine position after 10 minutes of rest. Higher values indicate increased arterial stiffness.
Ankle-Brachial Index (ABI) | From enrollment to the end of treatment at 12 weeks
  ABI is calculated as the ratio of the systolic blood pressure at the ankle (posterior tibial artery) to that in the arm (brachial artery), using a handheld Doppler ultrasound device. Measurements will be taken bilaterally (left and right sides), and the lower of the two values will be used for analysis.
  ABI values typically range from 0.00 to 2.00, with higher scores indicating better arterial perfusion.
  Values below 0.90 may indicate peripheral arterial disease (PAD), while values above 1.30 may suggest arterial stiffness or calcification.
Cardiorespiratory Fitness - Maximal Oxygen Uptake (VO2max) | From enrollment to the end of treatment at 12 weeks
  VO2max will be assessed via a graded exercise treadmill test using the Bruce protocol. Participants will wear a metabolic analyzer (e.g., Cortex MetaLyzer 3B) to measure oxygen consumption. The highest VO2 achieved before exhaustion will be recorded.
Peak Exercise Heart Rate (bpm) | From enrollment to the end of treatment at 12 weeks
  Heart rate at maximal effort during the Bruce treadmill test will be continuously monitored using a chest-worn heart rate monitor (e.g., Polar H10). The peak value during the test will be used for analysis.

OTHER OUTCOMES:
Weight | From enrollment to the end of treatment at 12 weeks
  Body weight will be measured using a calibrated digital scale with participants in light clothing, without shoes.Unit of Measure: Kilograms (kg).Higher values: May indicate weight gain; lower values may suggest weight loss.
Bone Mineral Density (BMD) | From enrollment to the end of treatment at 12 weeks
  BMD will be measured at the lumbar spine (L1-L4) and femoral neck using dual-energy X-ray absorptiometry (DXA; e.g., Hologic Discovery A). Results will be expressed as grams per square centimeter (g/cm²), representing the mineral density of bone tissue.Unit of Measure: g/cm².Higher values: Indicate better bone mineral density.
Body Mass Index (BMI) | From enrollment to the end of treatment at 12 weeks
  BMI will be calculated as weight in kilograms divided by the square of height in meters (kg/m²), using measured height and weight. It is a standard measure of body fatness.Unit of Measure: kg/m².Higher values: Indicate greater body mass.
Body Fat Percentage | From enrollment to the end of treatment at 12 weeks
  Body fat percentage will be assessed using dual-energy X-ray absorptiometry (DXA; e.g., Hologic Discovery A). It represents the proportion of fat to total body mass.Unit of Measure: Percent (%).Higher values: Indicate greater fat accumulation.
Fat Mass | From enrollment to the end of treatment at 12 weeks
  Fat mass will be measured using dual-energy X-ray absorptiometry (DXA; e.g., Hologic Discovery A). It represents the total weight of fat tissue in the body, excluding lean mass and bone. Participants will undergo DXA scanning in light clothing with all metal accessories removed.Unit of Measure: Kilograms (kg).
  Higher values: Indicate greater total fat accumulation.
Muscle Mass | From enrollment to the end of treatment at 12 weeks
  Muscle mass will be estimated using DXA (e.g., Hologic Discovery A), based on the sum of appendicular lean mass (four limbs). Results are reported in kilograms (converted from grams if necessary).Unit of Measure: Kilograms (kg).Higher values: Indicate greater muscle mass.
T-score | From enrollment to the end of treatment at 12 weeks
  T-score will be derived from DXA scans of the lumbar spine and femoral neck. It reflects the number of standard deviations by which the BMD differs from the mean of a healthy young adult reference population. T-score is used to diagnose osteopenia and osteoporosis.Unit of Measure: Unitless (Standard deviation, SD).Higher values: Indicate better bone status; values below -2.5 indicate osteoporosis.
Z-score | From enrollment to the end of treatment at 12 weeks
  Z-score will be derived from DXA scans and represents the number of standard deviations a participant's BMD is from the mean of age- and sex-matched controls.Unit of Measure: Unitless (Standard deviation, SD).Higher values: Indicate relatively better bone density for age.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The dataset will remain confidential in accordance with ethical and regulatory requirements to protect participant privacy.